CLINICAL TRIAL: NCT06113393
Title: Comparison of the Effects of Different Gastric Residual Volume Thresholds for Holding Enteral Feeding on Nutritional Intake in Critically Ill Patients in Internal Medicine
Brief Title: The Effects of Different Gastric Residual Volume Thresholds for Holding Feeding in Internal Medicine.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202307181RINB
Record Dates: First submitted 2023-10-22; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness
Keywords: Enteral nutrition; Gastric residual volume
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Hold enteral feeding when GRV reaches 200 mL(current standard)
- study group (Experimental): Hold enteral feeding when GRV reaches 300 mL(current standard)
  Interventions: Procedure: GRV thresholds

INTERVENTIONS:
Procedure: GRV thresholds — Hold enteral feeding when GRV reaches 200 mL(current standard)
  Arms: study group

SUMMARY:
This is a randomized control trial with a parallel design. Eligible patients will be randomly assigned into two groups: a control group which will be holding tube feeding when the GRV reaches 200 mL, and an experimental group will hold tube feeding when the GRV reaches 300 mL. Enteral feeding will be administered according to the study flow chart.

DETAILED DESCRIPTION:
Background: Malnutrition is a common issue among critically ill patients. which increases hospital stays, costs, and mortality rate. According to the study, the primary reason for nurses to hold enteral nutrition is elevated gastric residual volume (GRV). However, there is still no consensus on the definition of high residual gastric volume, there is currently no consensus among experts and scholars regarding the threshold for holding enteral nutrition. Clinical nurses may prematurely hold enteral nutrition due to concerns regarding potential side effects such as vomiting and choking. The aim of this study is to increase the threshold for holding enteral feeding based on the results of the study, in order to improve nutritional intake in critically ill patients in internal medicine.

Objective: Increase the nutritional intake of critically ill patients in the Department of Internal Medicine by increasing the threshold for holding tube feeding.

Methods: This is a randomized control trial with a parallel design. Eligible patients will be randomly assigned into two groups: a control group which will be holding tube feeding when the GRV reaches 200 mL, and an experimental group will hold tube feeding when the GRV reaches 300 mL. Enteral feeding will be administered according to the study flow chart. The outcome data will collected based on the medical chart including frequency of diet volume ratio (diet received/diet prescribed), incidence of gastrointestinal complications, ventilator days, Ventilator-associated pneumonia, length of intensive care unit(ICU) stay, changes in nutritional indicators, APACHE Ⅱ and Duration of parenteral nutrition use.

Expected result: The results of this study will provide evidence regarding the improved effectiveness and safety of increasing the threshold of GRV in medical ICU and inform future evidence-based practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the internal medicine intensive care unit.
* Patients receive enteral nutrition through a nasogastric tube.
* Patients receiving continuous enteral feeding.

Exclusion Criteria:

* Patients post-abdominal surgery.
* Patients admitted to the intensive care unit due to gastrointestinal disorders (e.g., gastrointestinal bleeding, bowel obstruction).
* Patients receiving palliative care with reduced enteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of diet volume ratio | 1 day (Transfer from the Intensive Care Unit)
Incidence of gastrointestinal complications | 1 day (Transfer from the Intensive Care Unit)
  Abdominal distension, nausea, vomiting, diarrhea, constipation

SECONDARY OUTCOMES:
Days of ventilator use | A week(Transfer from the Intensive Care Unit)
Ventilator-associated pneumonia | 1 day (Transfer from the Intensive Care Unit)
  Diagnosis form clinical doctor according to chest x-ray
Length of stay in the intensive care unit | A week(Transfer from the Intensive Care Unit)
Days of parenteral nutrition use | A week(Transfer from the Intensive Care Unit)
Acute Physiology and Chronic Health Evaluation score | 1 day (Transfer from the Intensive Care Unit)
  an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
Nutrition Risk Screening 2002(NRS2002) | 1 day (Transfer from the Intensive Care Unit)
  The NRS-2002 was developed by Kondrup et al., and is meant to be a generic tool in the hospital setting-that is, useful in detecting most of the patients who would benefit from nutritional therapy. The NRS-2002 is a simple and well-validated tool that incorporates pre-screening with four questions. If one of these is answered positively, a screening follows which includes surrogate measures of nutritional status, with static and dynamic parameters and data on the severity of the disease (stress metabolism). For each parameter, a score from 0 to 3 can result. Age over 70 years is considered a risk factor and is included in the screening tool, giving 1 point. A total score of ≥3 points means that the patient is at risk of malnutrition or already malnourished.
Albumin in g/dL | 1 day (Transfer from the Intensive Care Unit)
C-reactive protein in mg/dl | 1 day (Transfer from the Intensive Care Unit)
Body mass index | 1 day (Transfer from the Intensive Care Unit)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided